CLINICAL TRIAL: NCT03593577
Title: Saccular Dilatation, Endolymphatic Hydrops and Vestibular Schwannoma : is Vertigo Really Correlated to the Tumor ? A Retrospective Study Based on FIESTA-C Sequence Using a 3 Tesla MRI
Brief Title: Secondary Endolymphatic Hydrops and Vestibular Schwannomas on 3 Tesla MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7025
Record Dates: First submitted 2018-06-22; First posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-06

CONDITIONS: Vestibular Schwannoma
Keywords: Schwannoma; saccular dilatation; endolymphatic hydrops; magnetic resonnance imaging; vertigo
MeSH Terms: conditions — Neuroma, Acoustic; Neurilemmoma; Endolymphatic Hydrops; Vertigo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endolymphatic hydrops is well known of the lay public in its primary form that is Ménière disease. Nowadays, the best w ay to approach it in vivo, is to use magnetic resonance imaging (MRI).

However, endolymphatic hydrops don't limit itself to its primary form but cover a whole range of pathologies.

The hypothesis is that patients with vestibular schwannomas are more likely to develop secondary saccular hydrops.

The aim is to compare high-resolution T2-weighted images of the saccule in patients followed up for vestibular schwannomas with healthy volunteers and histological sections from cadavers in order to identify its changes.

The secondary purpose of The protocol is to determine if vestibular and audiometric abnormalities could be related to this secondary hydrops more specifically than to the tumor size and localisation.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18,
* Subject having benefited from an MRI with T2 high-resolution 3D sequence (FIESA) in the context of the diagnosis of vestibular schwannoma between 2008 and 2017 at the University Hospitals of Strasbourg,
* Subject who has agreed to the use of medical data for the purposes of this research.

Exclusion Criteria:

* Refusal of the patient to participate in the study
* Insufficient imaging data,
* Tumors already treated,
* Atypical tumors with uncertain diagnosis, intra-labrinthic or intra-labyrinthine schwannomas, concomitant infectious or inflammatory pathology in the middle or inner ear.
* Impossibility of giving the subject informed information (difficulty understanding the subject,)
* Subject under the protection of justice
* Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient having benefited from an MRI with T2 high-resolution 3D sequence (FIESA) in the context of the diagnosis of vestibular schwannoma between 2008 and 2017 at the University Hospitals of Strasbourg,
Sampling Method: Non-Probability Sample
Enrollment: 185 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of height and width of the saccule on MRI. | 1 hour after the realization of the MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Service Imagerie 1, Strasbourg, France